CLINICAL TRIAL: NCT00419354
Title: The Impact of Right Ventricular Pacing on Tricuspid Regurgitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Mordehay Vaturi/MD, Rabin Medical Center
Other Study IDs: 4134
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2006-07

CONDITIONS: Tricuspid Regurgitation
Keywords: Pacemaker; Tricuspid regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
"1" To examine whether right ventricular pacing has an impact on tricuspid regurgitation grade that is related to pacing rather than to valve closure interference by the electrode.

DETAILED DESCRIPTION:
"1" Traditionally, tricuspid regurgitation in the presence of pacemaker is attributed to the physical interference of the valve closure by the electrode.

"2" Right ventricular pacing may be associated with dyssynchrony in contraction of the right ventricular wall (i.e. septum and free wall.

"3" The tricuspid sub-valvar apparatus is anchored to the septum and free wall, thus may be sensitive to dyssynchrony in those wals contraction.

"4" The study hypothesis is that the dyssynchrony in right ventricular contraction, induced by pacing, may increase tricuspid regurgitation grade and that this is a mechanism is independent of the mechanical effect of the electrode on the valve closure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Permanent pacemaker

Exclusion Criteria:

* Epicardial pacing
* Left ventricular dysfunction
* Organic tricuspid regurgitation
* Bi-ventricular pacemaker
* Atrial fibrillation
* Complete pacemaker dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients, clinically stable, with a permanent pacemaker and who are not pacemaker dependent.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mordehay Vaturi, MD, Principal Investigator — Department of Cardiology, Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel